CLINICAL TRIAL: NCT05758740
Title: The Effectiveness of an E-health Brisk Walking Intervention in Increasing Moderate to Vigorous Physical Activity in Physically Inactive Older People With Cognitive Frailty: A Randomised Controlled Trial
Brief Title: E-health Brisk Walking in Older People With Cognitive Frailty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tung Wah College (Other)
Collaborators: The Hong Kong Polytechnic University (Other); University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UGC/FDS17/H04/22
Record Dates: First submitted 2023-02-13; First posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Cognitive Frailty
Keywords: e-health; brisk walking; moderate-to-vigorous physical activity; physical inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-health enhanced behavioural change intervention (Experimental): The investigators will administer e-health behavioural change techniques (e.g., automated advice, tele-counselling, digital-tailored advice) on top of the conventional behavioural change techniques (e.g., information provision, goal setting) via digital devices (i.e., smartphone) to promote moderate-to-vigorous physical activity of the participants.
  Interventions: Behavioral: E-health enhanced behavioural change intervention
- Conventional behavioural change intervention (Active Comparator): The investigators will administer conventional behavioural change techniques (e.g., information provision, goal setting) via conventional methods (i.e., face-to-face meetings) to promote moderate-to-vigorous physical activity of the participants.
  Interventions: Behavioral: Conventional behavioural change intervention

INTERVENTIONS:
Behavioral: E-health enhanced behavioural change intervention — Participants will first receive a face-to-face brisk-walking training programme with lectures and demonstrations following a standardized brisk training content. The training will be provided face-to-face at the elderly community centres and parks. Each training session lasts for one hour and is two times per week for two weeks. After that, a conventional behavioural change intervention will begin following a standardized intervention implementation manual and the physical activity amount will be logged by the participants using a logbook. Physical activity counselling will be conducted by a trained research assistant face-to-face at the elderly community centre. Each counselling session lasts for one hour and is once per week for 12 weeks.
  Arms: E-health enhanced behavioural change intervention
Behavioral: Conventional behavioural change intervention — Participants will first receive a face-to-face brisk-walking training programme with lectures and demonstrations following a standardized brisk training content. The training will be provided face-to-face at the elderly community centres and parks. Each training session lasts for one hour and is two times per week for two weeks. After that, e-health enhanced behavioural change intervention will begin following a standardized intervention implementation manual and using participants' own smartphones installed with two Apps (i.e., Samsung Health and WhatsApp). The physical activity amount will be logged by the smartphone using Samsung Health. Physical activity counselling will be conducted by a trained research assistant remotely using a smartphone. The remote counselling sessions totally last for accumulatively 1 hour per week for 12 weeks.
  Arms: Conventional behavioural change intervention

SUMMARY:
Introduction Cognitive frailty is common in community-dwelling older people and is an at-risk state for adverse health outcomes such as dementia, dependency, and mortality. Fortunately, cognitive frailty is reversible, with a higher probability of reversibility at earlier stages. Physical activity is known to play a significant role in reversing cognitive frailty; its effect is moderated by intensity and sustainability. However, physical inactivity is very common in older people and is one of the key phenotypical characteristics of cognitive frailty. Moderate to vigorous physical activity (MVPA) can reduce the risk of worsening cognitive frailty. Brisk walking is a simple form of exercise that can be practised by community-dwelling older people every day to boost their physical activity to or above a moderate intensity level. Conventional behavioural change interventions (CBCIs) have been shown to effectively engage sedentary older people in physical activity, but their effect size is small. The use of e-health methods that adopt existing and popular e-platforms (e.g., Samsung Health and WhatsApp) to promote specific behaviours (e.g., regular brisk walking) in specific groups (e.g., older people with cognitive frailty) is an innovative, practically feasible and theoretically sound method of increasing MVPA. However, the relative effectiveness of e-health interventions and CBCIs in vulnerable groups (i.e., older people with cognitive frailty) is unknown.

Objectives The objectives of this study are to compare the effectiveness of an e-health intervention and a conventional behavioural change intervention in older people with cognitive frailty in improving 1) moderate-to-vigorous physical activity, 2) reducing cognitive frailty, 3) improving cognitive function, 4) improving walking speed, 5) improving functional fitness, and 6) improving physical activity motivation

Methods A single-blinded, two-parallel-group, non-inferiority, randomised controlled trial will be conducted in a community setting. Subjects will be recruited from five elderly community centres in Hong Kong. The eligibility criteria will be as follows: (1) aged ≥ 60, (2) cognitively frail, (3) physically inactive and (4) possessing a smartphone. The participants in the intervention group will receive an e-health intervention. Those in the control group will receive a CBCI. Each intervention will last for 14 weeks. The outcomes will be MVPA min/week (primary), as measured by a wrist-worn ActiGraph; cognitive frailty, as measured by an ordinal scale; cognitive function, as measured by the Montreal Cognitive Assessment; and frailty, as measured by the Fried frailty phenotype (FFP). The outcomes will be assessed at T0 (baseline), T1 (immediately post-intervention) and T2 (6 months post-intervention). The investigators plan to recruit 192 subjects. Permuted block randomisation with randomly selected block sizes in a ratio of 1:1 will be used. Only the outcome assessors will be blinded. Four generalised estimating equations will be used to test the effects of the interventions on the four outcomes, which will be the dependent variables. The independent variables will be group, time and [group] × [time]. The level of significance will be set at 0.05.

Significance If the e-health intervention proves to be more effective and sustainable than the CBCI, There will be evidence suggesting that e-health interventions can replace CBCIs in promoting MVPA and treating cognitive frailty in older people in community settings. Further studies could then examine the potential role of e-health interventions in delaying the onset of dementia and dependency.

ELIGIBILITY:
Inclusion Criteria:

* 1) aged ≥ 60 years, because the WHO defines older people in Asia as those aged 60 or older;
* 2) presence of cognitive frailty, defined as the co-existence of MCI and frailty at either the pre-frail or the frail level;
* 3) physical inactivity, defined as < 150 min of MVPA every week in the 4 weeks preceding the study, as confirmed by a Rapid Assessment of Physical Activity (RAPA) score of ≤ 4 (i.e., regularly underactive);
* 4) possession of a smartphone on which Samsung Health and WhatsApp can be installed for > 6 months; and
* 5) being a Cantonese speaker, defined as possessing the ability to communicate in Cantonese.

Exclusion Criteria:

* 1) impaired mobility caused by conditions that require medication (e.g., severe arthritis) and inability to walk briskly outdoors, as defined by a modified Functional Ambulatory Classification score of < 7);
* 2) depressive symptomatology, as defined by a Geriatric Depression Scale (GDS) score of ≥ 8;67
* 3) having probable dementia (i.e., a Montreal Cognitive Assessment [MoCA] score of < 20 or Clinical Dementia Rating [CDR] score of ≥ 1),
* 4) being physically unfit because of chronic illness, as defined by a Physical Activity Readiness Questionnaire (PAR-Q) score of ≥ 1, and not having been examined by a medical doctor and certified as physically fit to participate in brisk walking;
* 5) not enrolled in any other interventions to promote physical activity or training

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Moderate-to-vigorous physical activity (MVPA) minute, measured by Actigraph | 14 weeks
  ActiGraph mounted on the right wrist measures physical movement (i.e., vector magnitude) that counts an MVPA minute when it has measured 4,212.9 counts within a minute. Only at least 10 min of continuous MVPA will be counted as valid MVPA minutes. This variable measures valid MVPA minutes accumulated over 7 consecutive days.
Moderate-to-vigorous physical activity (MVPA) minute, measured by Actigraph | 6 months
  ActiGraph mounted on the right wrist measures physical movement (i.e., vector magnitude) that counts an MVPA minute when it has measured 4,212.9 counts within a minute. Only at least 10 min of continuous MVPA will be counted as valid MVPA minutes. This variable measures valid MVPA minutes accumulated over 7 consecutive days.

SECONDARY OUTCOMES:
Cognitive frailty, measured by a 6-point scale of Cognitive Frailty | 14 weeks
  Cognitive frailty comprises six combinations of two components: frailty (robust, pre-frail, and frail) and mild cognitive impairment (yes, no). The scale quantifies cognitive frailty at six levels: 0 for "robust without mild cognitive impairment", 1 for "pre-frail without mild cognitive impairment", 2 for "frail without mild cognitive impairment", 3 for "non-frail with mild cognitive impairment", 4 for "pre-frail with mild cognitive impairment" and 5 for "frailty with mild cognitive impairment". A higher score will indicate greater severity of cognitive frailty.
Cognitive frailty, measured by a 6-point scale of Cognitive Frailty | 6 months
  Cognitive frailty comprises six combinations of two components: frailty (robust, pre-frail, and frail) and mild cognitive impairment (yes, no). The scale quantifies cognitive frailty at six levels: 0 for "robust without mild cognitive impairment", 1 for "pre-frail without mild cognitive impairment", 2 for "frail without mild cognitive impairment", 3 for "non-frail with mild cognitive impairment", 4 for "pre-frail with mild cognitive impairment" and 5 for "frailty with mild cognitive impairment". A higher score will indicate greater severity of cognitive frailty.
Cognitive function, measured by Montreal Cognitive Assessment | 14 weeks
  Montreal Cognitive Assessment comprises 30 dichotomous items. One point will be assigned to one correct answer. The total score ranges from 0 to 30. A higher score indicates a higher level of cognitive function.
Cognitive function, measured by Montreal Cognitive Assessment | 6 months
  Montreal Cognitive Assessment comprises 30 dichotomous items. One point will be assigned to one correct answer. The total score ranges from 0 to 30. A higher score indicates a higher level of cognitive function.
Walking speed, measured by Timed Up-and-Go Test | 14 weeks
  Timed Up-and-Go test measures the total time needed for a participant to stand up from a chair, walk a 3-metre distance, walk back to the chair, and sit down. A longer time needed to complete the test indicates a slower walking speed.
Walking speed, measured by Timed Up-and-Go Test | 6 months
  Timed Up-and-Go test measures the total time needed for a participant to stand up from a chair, walk a 3-metre distance, walk back to the chair, and sit down. A longer time needed to complete the test indicates a slower walking speed.
Functional fitness, measured by 30-second Chair Stand Test | 14 weeks
  30-second Chair Stand Test measures the number of stands a person can complete in 30 seconds. A higher number of stands completed within the given 30 seconds indicates a higher level of functional fitness.
Functional fitness, measured by 30-second Chair Stand Test | 6 months
  30-second Chair Stand Test measures the number of stands a person can complete in 30 seconds. A higher number of stands completed within the given 30 seconds indicates a higher level of functional fitness.
Physical activity motivation, measured by Revised Motivation for Physical Activity Measure | 14 weeks
  Revised Motivation for Physical Activity Measure comprises 30 7-point items with a total score ranging from 30 to 210. A higher score indicates greater motivation to perform physical activity.
Physical activity motivation, measured by Revised Motivation for Physical Activity Measure | 6 months
  Revised Motivation for Physical Activity Measure comprises 30 7-point items with a total score ranging from 30 to 210. A higher score indicates greater motivation to perform physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Rick Kwan, PhD, Principal Investigator — School of Nursing, Tung Wah College

IPD SHARING:
Plan to Share IPD: Undecided
Data will be provided upon other researchers' requests

REFERENCES:
- [Derived] Kwan RYC, Liu JYW, Lee PH, Sin OSK, Wong JSW, Fu MR, Suen LKP. The effects of an e-health brisk walking intervention in increasing moderate-to-vigorous physical activity in physically inactive older people with cognitive frailty: study protocol for a randomized controlled trial. Trials. 2023 May 17;24(1):339. doi: 10.1186/s13063-023-07335-8. PMID 37198670